CLINICAL TRIAL: NCT03953378
Title: Presence and Impact of CD73+ Th1.17 and of the CD39/CD73/Adenosine Cascade in Rheumatoid Arthritis (RA) and Psoriatic Arthritis (PsA)
Brief Title: CD73+ Th1.17 in Rheumatoid Arthritis and Psoriatic Arthritis
Acronym: LAdoRIC
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: LAdoRIC
Record Dates: First submitted 2019-05-13; First posted 2019-05-16 (Actual); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Rheumatoid Arthritis; Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group "RA patients": Patients with Rheumatoid Arthritis (RA) fulfilling the American College of Rheumatology and European League Against Rheumatism 2009 criteria.
  Interventions: Other: Multi-parametric Flow Cytometry analysis on patients and healthy donors samples
- Group "PsA patients": Patients with Psoriatic Arthritis (PsA) fulfilling the Classification for PsA (CASPAR) criteria.
  Interventions: Other: Multi-parametric Flow Cytometry analysis on patients and healthy donors samples
- Group "Healthy donors": Anonymous healthy donors from the Etablissement Français du Sang.
  Interventions: Other: Multi-parametric Flow Cytometry analysis on patients and healthy donors samples

INTERVENTIONS:
Other: Multi-parametric Flow Cytometry analysis on patients and healthy donors samples — Collection of venous blood (16 mL) and synovial fluid (when available) samples, for each patient, at inclusion and in the frame of the usual medical follow-up at 3 months and between 6 and 12 months, before the onset of MTX (untreated patients) or during the course of MTX treatment (MTX-treated patients).
  Collection of anonymous healthy donors blood samples, age- and sex-matched, obtained from the Etablissement Français du Sang.
  Multi-parametric Flow Cytometry analysis was performed on these samples to assess CD73 expression on total memory T cells and within T helper lymphocyte subsets, their cytokine production and AMPase functions. For FoxP3 intracellular staining, cells were treated using the FoxP3 Fixation and Permeabilization kit (Life Technologies), according to manufacturer instructions. Stainings were analyzed on a LSR-Fortessa™ (BD Biosciences) with conserved settings throughout the entire study and data were analyzed using FlowJo™ Software (Tree Star v10.4).

SUMMARY:
Prospective study to investigate the correlation between CD39/CD73 expression by the different T lymphocyte subpopulations in the blood and synovial fluid (if available) into patients with chronic inflammatory rheumatism RA and PsA types, with the rheumatic activity, the background therapy (with Methotrexate (MTX)) and the response to this treatment.

DETAILED DESCRIPTION:
Th1.17 compose a recently described subset of highly polyfunctional and thus potentially more harmful CD4+ effector T cells (Teff) than classical Th17 as they co-produce interferon-γ (IFN-γ) and interleukin-17A (IL-17A). For this reason, Th1.17 rise increasing interest in RA and PsA since they seem involved in their pathophysiology. Hyper activation of Teff in RA and PsA results partly from a deficiency in regulatory mechanisms of Teff's pro-inflammatory functions. The ecto-nucleotidase CD73 delineates Teff enriched in Th1.17 features and acts as a regulatory mechanism for these pro-inflammatory cells. Considering that MTX, usually used as first line treatment of RA and PsA, increases extracellular concentrations of adenosine monophasphate (AMP) and immunosuppressive adenosine, the investigators hypothesized that CD4+CD73+ T cell effector population enriched in Th1.17 and Th17 cells may participate in the pathogenicity of RA and PsA but also in the resistance to MTX treatment through the specific expression of CD73 essential for Ado generation and which is down-regulated on proliferating T cells.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years
* Patients naive to biologics
* Patients with RA fulfilling the American College of Rheumatology and European League Against Rheumatism 2009 criteria
* Patients with PsA fulfilling the Classification for PsA (CASPAR) criteria

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic inflammatory rheumatism RA and PsA types with or without background therapy at the inclsuion
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
CD73 expression on T helper lymphocyte subpopulations | At inclusion
  Determine CD73 expression on T helper lymphocyte subpopulations (using multi-parametric Flow Cytometry), in the blood and synovial fluid of Rheumatoid Arthritis (RA) or Psoriatic Arthritis (PsA) patients before or under MTX treatment.
CD73 expression on T helper lymphocyte subpopulations | 3 months
  Determine CD73 expression on T helper lymphocyte subpopulations (using multi-parametric Flow Cytometry), in the blood and synovial fluid of Rheumatoid Arthritis (RA) or Psoriatic Arthritis (PsA) patients before or under MTX treatment.
CD73 expression on T helper lymphocyte subpopulations | 12 months
  Determine CD73 expression on T helper lymphocyte subpopulations (using multi-parametric Flow Cytometry), in the blood and synovial fluid of Rheumatoid Arthritis (RA) or Psoriatic Arthritis (PsA) patients before or under MTX treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Rhumatologie, Centre Hospitalier Lyon-Sud (HCL), Pierre-Bénite, France